CLINICAL TRIAL: NCT06184217
Title: Effects of the Mindfulness Sport Performance Enhancement Programme on Competitive Athletes With Physical Disabilities.
Brief Title: Effects of a Mindfulness Programme on Competitive Athletes With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Sandra Constantino Murillo, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPM
Record Dates: First submitted 2023-11-26; First posted 2023-12-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Athletic Injuries; Physical Disability; Chronic Pain
Keywords: Athlete Injuries; Physical disability; Chronic pain; Psychological abilities; Mindfulness
MeSH Terms: conditions — Athletic Injuries; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (MSPE programme group). (Experimental): Experimental (MSPE group). The experimental group received the Mindful Sport Performance Enhancement programme (MSPE), with some changes and adaptations taking into account the characteristics and needs of the Para-athletes and the overall aim of the study. Such as reducing the session time (2h), including staff and support material, extending the pre-session time (35-40 min), and incorporating the dynamics of emotions and Mindful Yoga into the floor of the MBSR programme [2].
  Interventions: Other: Experimental group (MSPE programme group).
- Control group (relaxation group). (Active Comparator): Control group. Control group. Athletes with physical disabilities participating in the home were provided with a guide to body awareness-based relaxation training guidelines [3].
  Interventions: Other: Control group (relaxation group).

INTERVENTIONS:
Other: Experimental group (MSPE programme group). — Experimental group. MSPE Programme. This group will receive a face-to-face mindfulness MSPE programme for 6 weeks, once a week for 1h 50min-2 hours. In addition to doing mindfulness activities at home. Each session contains the following exercises: (1) intention meditation, sultana exercise, diaphragmatic breathing and sitting meditation with a focus on breath, body and sound; (2) diaphragmatic breathing, Body Scan; (3) sitting meditation, dynamics of emotions, Mindful Yoga on the floor; (4) letting go of attachments, mindful Yoga on the floor walking meditation; (5) sports meditation, sitting meditation with a focus on breath, body and sound; (6) intention meditation, body scan analysis and review of sports meditation.
  Arms: Experimental group (MSPE programme group).
Other: Control group (relaxation group). — These instructions included a combination of tension-relaxation of specific muscles and simple breathing techniques. They were recommended to do this on a daily basis, with a minimum of 4 sessions per week.
  Arms: Control group (relaxation group).

SUMMARY:
Pain affects the athlete's sporting career directly or indirectly. Directly, the injury affects other areas of the body causing a physical decompensation in the athlete and this affects the correct execution of the sporting technique, or how technical gestures can cause pain. Indirectly, through the psychological consequences of pain that generate a series of negative consequences and feelings. Some studies suggest that psychological skills are an important tool for pain management. For that reason, a mindfulness intervention programme would be a useful tool for manage pain in this population.

DETAILED DESCRIPTION:
The study hypothesised that the Mindfulness Sports Performance Enhancement (MSPE) programme adapted for this population, was more effective than mindfulness-based relaxation training as a treatment for chronic pain and associated emotional disturbances in Para athletes with physical disabilities, and that it contributes more to modifying psychological variables that have been shown to be related to or have modulatory value in the experience of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a physical disability
* A minimum of 5 points on a Likert-type scale from 1 (no pain) to 10 (worst pain imaginable) at the time of recruitment
* Be at least 15 years of age
* Have been a competitive athlete (regional, national, world and/or Paralympic Games level) in any sport discipline.
* Have an official regional or Spanish Federation of Sports for People with Physical disabilities licence
* Be willing to participate in a mindfulness programme for pain management
* Sign an informed consent form.

Exclusion Criteria:

* Not having at least one of the criteria mentioned as inclusion.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (current pain) post intervention. [Time Frame: Baseline and at 6 weeks].[Safety Issue: No]. | Month and a half.
  The presence of pain intensity (current pain) will be measured on a visual analogue Likert-type rating scale from 1 (no pain) to 10 (worst pain imaginable) without and with sports practice. A higher score indicates greater intensity.
Change in pain frequency post intervention. [Time Frame: Baseline and at 6 weeks].[Safety Issue: No] | Month and a half.
  The frequency with which Para-athletes experience pain will be assessed on a Likert-type scale from 1 (very infrequent) to 5 (very frequent).

SECONDARY OUTCOMES:
Secondary Outcome Measure. [Time Frame: Baseline and at 6 weeks].[Safety Issue: No]. Higher values reflect higher levels on the scale to be measured. | Month and a half.
  Mindfulness: 2. Mindful Attention Awareness Scale (MAAS). The scale will assess the individual's ability to be attentive and aware of the present moment experience in everyday life. ID: 22344492.
  Mental health variables:
  3. Depression, Anxiety, and Stress Scales (DASS-21). The scale will assess the presence and intensity of affective states of depression, anxiety, and stress. [5].
  4. Scales of Psychological Well-Being (SPWBP). The scale will assess the six dimensions postulated in the multidimensional model of psychological well-being. ID de PubMed: 17296089.
  5. Satisfaction with Life Scale (SWLS). The scale will assess satisfaction with life. [7].
  Coping strategies:
  6. Chronic Pain Acceptance Questionnaire (CPAQ). This questionnaire measures involvement in activities and openness to pain. ID: 21044544.
  7. Coping Strategies Questionnaire (CSQ). This questionnaire will assess the frequency with which the subject uses different pain coping strategies. ID: 15042468

CONTACTS AND LOCATIONS:
Overall Officials: María I. B Barriopedro, PhD in Psychology, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Sandra Constantino Murillo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [1] Kaufman, K., Glass, C. R., & Pineau, T. R. (2018). Mindful sport performance enhancement: Mental training for athletes and coaches. American Psychological Association.
- [Background] [2] Martín-Asuero (2008). On your own course. Enjoy life without stress. Platform.
- [Background] [3] Bernstein, D., Borkovec, T., & Hazlett-Stevens, H. (2000). New Directions in Progressive Relaxation Training: A Guidebook for Helping Professionals. Bloomsbury Academic.
- [Background] Soler J, Tejedor R, Feliu-Soler A, Pascual JC, Cebolla A, Soriano J, Alvarez E, Perez V. Psychometric proprieties of Spanish version of Mindful Attention Awareness Scale (MAAS). Actas Esp Psiquiatr. 2012 Jan-Feb;40(1):19-26. Epub 2012 Jan 1. PMID 22344492
- [Background] [5] Daza P, Novy DM, Stanley MA, Averill P. The depression, anxiety, stress-21 scale: translation and validation into Spanish with a Hispanic sample. Journal of Psychopathology and Behavioral Assessment. 2002; 24(3): 195-205.
- [Background] Diaz D, Rodriguez-Carvajal R, Blanco A, Moreno-Jimenez B, Gallardo I, Valle C, van Dierendonck D. [Spanish adaptation of the Psychological Well-Being Scales (PWBS)]. Psicothema. 2006 Aug;18(3):572-7. Spanish. PMID 17296089
- [Background] Pons D, Atienza FL, Balaguer I, Garcia-Merita ML. Satisfaction with life scale: analysis of factorial invariance for adolescents and elderly persons. Percept Mot Skills. 2000 Aug;91(1):62-8. doi: 10.2466/pms.2000.91.1.62. PMID 11011872
- [Background] Gonzalez Menendez A, Fernandez Garcia P, Torres Viejo I. [Acceptance of chronic pain in fibromyalgia patients: adaptation of Chronic Pain Acceptance Questionnaire (CPAQ) in a Spanish population]. Psicothema. 2010 Nov;22(4):997-1003. Spanish. PMID 21044544
- [Background] Rodriguez Franco L, Cano Garcia FJ, Blanco Picabia A. [Assessment of chronic pain coping strategies]. Actas Esp Psiquiatr. 2004 Mar-Apr;32(2):82-91. Spanish. PMID 15042468